CLINICAL TRIAL: NCT03784716
Title: Ke-To Liver Health Study: A Randomized Controlled Trial to Study the Effects of a 28-day Ketogenic Dietary Intervention on Non-alcoholic Fatty Liver Disease Progression
Brief Title: Ketogenic Diet in Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marc Goodman (Other)
Responsible Party: Sponsor-Investigator, Marc Goodman, Principal Investigator; Director Cancer Prevention and Control; Professor, Department Cancer Institute, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2018-27-Hussain-KetoLi
Record Dates: First submitted 2018-12-04; First posted 2018-12-24 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Fatty Liver, Nonalcoholic; Liver Diseases
Keywords: Fatty Liver; Liver Disease; Ketogenic diet; Keto diet
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases; Fatty Liver | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic Diet (Experimental): Ketogenic Diet for 28 Days
  Interventions: Other: Ketogenic Diet
- Standard Weight Loss Diet (Active Comparator): Standard Weight Loss Diet for 28 Days
  Interventions: Other: Standard Weight Loss Diet

INTERVENTIONS:
Other: Ketogenic Diet — Ketogenic diet for 28 days. Meals will be provided to all study participants for 28 days by a prepared meal delivery service. Daily caloric needs for each participant will be determined based on height, weight, gender, age, and activity level. Meals will be prepared based on compliance with the following macronutrient guidelines: 70% fat, 25% protein, and 5% carbohydrate for the ketogenic diet.
  Arms: Ketogenic Diet
Other: Standard Weight Loss Diet — Standard weight loss diet for 28 days. Meals will be provided to all study participants for 28 days by a prepared meal delivery service. Daily caloric needs for each participant will be determined based on height, weight, gender, age, and activity level. Meals will be prepared based on compliance with the following macronutrient guidelines: 30% fat, 20% protein, and 50% carbohydrate for the standard weight loss diet.
  Arms: Standard Weight Loss Diet

SUMMARY:
The purpose of this randomized trial is to examine the effects of a ketogenic diet on non-alcoholic fatty liver disease (NAFLD). Twenty-four participants with NAFLD will be randomized to receive a ketogenic meal plan or control (standard weight loss meal plan). Participants will be followed up to 28 days after initiation of the diet intervention.

DETAILED DESCRIPTION:
We will conduct a randomized trial to examine the effects of a ketogenic diet on non-alcoholic fatty liver disease (NAFLD). Twenty-four participants with NAFLD will be randomized into one of two groups: 12 participants will be randomized to receive a ketogenic meal plan and 12 participants will be randomized to receive a standard weight loss meal plan. There will be one screening visit and three study visits: the baseline visit, and follow-up visits 14 days and 28 days after initiation of the diet intervention. The study team hypothesizes that participants randomized to a ketogenic diet will have a greater reduction in intrahepatic triglycerides compared to those randomized to a standard weight loss diet.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years at enrollment
* Diagnosis of NAFLD verified by screening MRI-PDFF greater than or equal to 8%
* Women able to become pregnant must have a confirmed negative pregnancy test result prior to enrollment because MRI is contraindicated in pregnant women. Women ≥ 50 years of age who have not had a menstrual period in the past year; and women who have had a hysterectomy, both ovaries removed, or a tubal ligation; will not be required to have a pregnancy test.
* Women able to become pregnant must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document and medical release
* Willing and able to comply with trial protocol and follow-up

Exclusion Criteria:

* Prior diagnosis of chronic liver disease other than NAFLD, including autoimmune, viral, and alcoholic liver disease
* Prior diagnosis of liver cirrhosis as defined by any of the following criteria:

  * Cirrhosis on historical liver biopsy; or
  * Evidence of cirrhosis on liver imaging (CT, MRI, or US) including a nodular liver surface, splenomegaly, or portal venous collaterals; or
  * Prior history of decompensated liver disease, including ascites, hepatic encephalopathy, or variceal bleeding; or
  * FibroScan value of >14.9 kPa; or
  * MRE of 4.67 kPa or higher
* History of liver transplantation
* Body mass index (BMI) less than 27 kg/m
* Unstable body weight (> 10% change in prior 3 months)
* Prior weight reduction surgery within the last 5 years
* Use of a medication prescribed for weight loss within the past 3 months
* Current alcohol consumption >21 oz. per week for males or >14 oz. per week for females (1 oz./30 mL of alcohol is present in one 12 oz./360 mL beer, one 4 oz./120 mL glass of wine, and one 1 oz./30 mL measure of 40% proof alcohol)
* Unstable cardiovascular disease as defined by any of the following:

  * Unstable angina within 6 months prior to screening
  * Myocardial infarction, coronary artery bypass graft surgery or coronary angioplasty within 6 months prior to screening
  * Transient ischemic attack or cerebrovascular accident within 6 months prior to screening
  * Obstructive valvular heart disease or hypertrophic cardiomyopathy
  * Unstable congestive heart failure
* Women who are pregnant or breastfeeding or are implanted with intrauterine devices that are not MRI-compatible
* Active malignancy within the past 5 years (excluding basal/squamous cell skin cancer, or prostate cancer with a Gleason score 6 or less)
* Known HIV infection
* Food allergies or dietary restrictions, including vegan or vegetarian diet, which cannot be accommodated with the prepared meal service
* Contraindication to undergo MRI-PDFF or MRE, including persons with mechanically, magnetically, or electrically activated implants, such as cardiac pacemakers or defibrillators, or infusion pumps; or ferromagnetic implants or foreign bodies, such as aneurysm clips or shrapnel; or other implanted electronic devices or metallic parts in the body prohibiting MRI. Because the MRI scanner is also used with animals, persons with allergy to animal dander or animal-instigated asthma are also excluded.
* Resides outside of the meal delivery zone or plans to travel outside of the meal delivery zone for more than one day while on the study intervention and will be unable to access the meal delivery
* Current use of any investigational agents
* Concurrent illness or abnormal laboratory result which in the opinion of the investigators would compromise either the patient or the integrity of the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Mean change in intrahepatic triglyceride content measured by MRI-proton density fat fraction (MRI-PDFF) from baseline to 28 days following diet initiation. | 28 days
  The MRI-PDFF is a quantitative imaging test that exploits the differences in resonance frequencies between

SECONDARY OUTCOMES:
Mean change in liver stiffness measured by magnetic resonance elastography (MRE) from baseline to 28 days following diet initiation. | 28 days
  Stiffness will be measured by MRE (kPa), a quantitative imaging test that uses sound vibrations to assess the mechanical properties of the liver.
Mean change in liver enzyme, aspertate aminotransferase (AST), from baseline to 28 days following diet initiation. | 28 days
  AST will be measured from blood test at baseline and 28 days from diet initiation
Mean change in liver enzyme, Alanine Aminotransferase (ALT), from baseline to 28 days following diet initiation. | 28 days
  ALT will be measured from blood test at baseline and 28 days from diet initiation
Mean change in number of odors correctly identified using 40 microencapsulated odors in the smell identification test (UPSIT) from baseline to 28 days following diet initiation. | 28 days
  The University of Pennsylvania Smell IdentificationTest (UPSIT) uses 40 microencapsulated odors embedded in questionnaire accompanied by multiple choice questions containing the correct odor.
Mean change in perceived sweet taste tested with glucose solutions and a general Labeled Magnitude Scale (gLMS) from baseline to 28 days following diet initiation. | 28 days
  Sweet taste intensity will be rated on a 100mm general Labeled Magnitude Scale (gLMS) ranging from no sensation (0 mm) to strongest imaginable sensation (100 mm). The mean difference in scores will be calculated at 28 days following diet initiation and baseline.
Mean change in patient-reported cognitive function measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) scale from baseline to 28 days following diet initiation. | 28 days
  Cognitive function will be assessed using the NIH Patient-Reported Outcomes Measurement Information System (PROMIS) short form, which includes 8 items and a range of 1 to 5 (worst outcome). The total score will be calculated and converted into a standardized t-score will be calculated based on a standard population with a mean of 50 and SD of 10.
Mean change in patient-reported constipation measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) scale from baseline to 28 days following diet initiation. | 28 days
  Constipation will be assessed using the NIH Patient-Reported Outcomes Measurement Information System (PROMIS) short form, which includes 9 items and a range of 1 (low constipation) to 5 (high constipation). The total score will be calculated and converted into a standardized t-score will be calculated based on a standard population with a mean of 50 and SD of 10.
Mean change in patient-reported fatigue measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) scale from baseline to 28 days following diet initiation. | 28 days
  Fatigue will be assessed using the NIH Patient-Reported Outcomes Measurement Information System (PROMIS) short form, which includes 8 items and a range of 1 (low fatigue) to 5 (high fatigue). The total score will be calculated and converted into a standardized t-score will be calculated based on a standard population with a mean of 50 and SD of 10.
Mean change in physical activity measured by a wearable activity monitor from baseline to 28 days following diet initiation. | 28 days
  A 7-day average at 28 days will be compared to 7-day baseline activity where at least 4 of 7 days of recorded activity required.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Goodman, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States